CLINICAL TRIAL: NCT01434589
Title: Effects of a Manualized Short-term Treatment of Internet and Computer Game Addiction
Acronym: STICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, M.E. Beutel, Univ.-Prof. Dr.med. Dipl.-Psych. M.E. Beutel, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BE 2248/10-1
Record Dates: First submitted 2011-09-08; First posted 2011-09-15 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Addiction
Keywords: internet addiction; computer game addiction; STICA; short-term treatment; psychotherapy; internet and computer game addiction
MeSH Terms: conditions — Behavior, Addictive; Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait list control (No Intervention)
- STICA Intervention (Experimental)
  Interventions: Behavioral: STICA Intervention

INTERVENTIONS:
Behavioral: STICA Intervention — Manualized Short-term Treatment for Internet and Computer game Addiction (STICA) based on cognitive behavior-therapy (combining individual and group therapy)
  Arms: STICA Intervention

SUMMARY:
The purpose of this study is to 1) determine the efficacy of manualized Short-term Treatment of Internet and Computer game Addiction (STICA), assess 2) the durability of treatment response in these patients and 3) the impact on associated psychiatric symptoms, e.g. social anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of internet or computer game addiction
* internet or computer game addiction according to the AICA-Checklist(Assessment of Internet and Computer game addiction, expert Rating)
* a score >/= 7 in the AICA-S (Assessment of Internet and Computer game addiction, Self Rating)
* patients with primary diagnoses of internet or computer game addiction
* if currently on psychotropic medications, no change in medications and dosages in the past 2 months and during STICA treatment
* if currently off all psychotropic medications, patient has been off at least 4 weeks
* at least 4 weeks off from last psychotherapy and no other ongoing psychotherapy

Exclusion Criteria:

* current Global Assessment of Functioning (GAF) < 40
* severe major depression (BDI-II Score >/= 29)
* current alcohol or drug addictions
* personality disorders: borderline, antisocial, schizoid and schizotypal
* lifetime diagnoses of schizophrenia, schizoaffective, bipolar or organic mental disorder
* current unstable medical illness

Ages: 17 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 187 (Actual)
Dates: Start 2012-01; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in internet or computer game addiction (self-rating) | 4 and 10 months after randomization

SECONDARY OUTCOMES:
Change/Remission of internet or computer game addiction (expert rating) | 4 and 10 months after randomization
Preoccupation with critical internet applications or computer games (hours per week) | 4 and 10 months after randomization
Improvement of negative consequences (e.g. social communication, psychosocial well being) | 4 and 10 months after randomization
Improvement of depressive symptoms (changes in BDI-II) | 4 and 10 months after randomization
Improvement of social fear and avoidance (changes in Liebowitz Social Anxiety Scale) | 4 and 10 months after randomization
Improvement of Expectances of self-efficacy (Changes in Assessment of Self-Efficacy) | 4 and 10 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: M. E. Beutel, Prof. Dr., Principal Investigator — University Medical Center Mainz, Department of Psychosomatic Medicine and Psychotherapy
Locations (4):
- Anton Proksch Insitut, Therapy Centre for the Treatment of Addictions, Vienna, Austria
- Germany (3):
  - University Medical Center Mainz, Department of Psychosomatic Medicine and Psychotherapy, Outpatient clinic for behavioral addictions, Mainz
  - Central Insitute for Mental Health, Mannheim
  - University Medical Center Tübingen, Tübingen

REFERENCES:
- [Background] Wolfling K, Muller KW, Beutel M. [Reliability and validity of the Scale for the Assessment of Pathological Computer-Gaming (CSV-S)]. Psychother Psychosom Med Psychol. 2011 May;61(5):216-24. doi: 10.1055/s-0030-1263145. Epub 2010 Sep 27. German. PMID 20878599
- [Derived] Wolfling K, Muller KW, Dreier M, Ruckes C, Deuster O, Batra A, Mann K, Musalek M, Schuster A, Lemenager T, Hanke S, Beutel ME. Efficacy of Short-term Treatment of Internet and Computer Game Addiction: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Oct 1;76(10):1018-1025. doi: 10.1001/jamapsychiatry.2019.1676. PMID 31290948
- [Derived] Jager S, Muller KW, Ruckes C, Wittig T, Batra A, Musalek M, Mann K, Wolfling K, Beutel ME. Effects of a manualized short-term treatment of internet and computer game addiction (STICA): study protocol for a randomized controlled trial. Trials. 2012 Apr 27;13:43. doi: 10.1186/1745-6215-13-43. PMID 22540330